CLINICAL TRIAL: NCT02920996
Title: A Phase II Study of Merestinib in Non-Small Cell Lung Cancers Harboring MET Exon 14 Mutations and Solid Tumors With NTRK Rearrangements
Brief Title: Merestinib In Non-Small Cell Lung Cancer And Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was pulled
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Mark Awad, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-374; I30-MC-E001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Solid Tumor
Keywords: NSCLC; MET; Non-small cell lung cancer; MET mutation; NTRK rearrangement; NTRK; targeted therapy; MET exon 14; NTRK1; NTRK2; NTRK3; merestinib; LY2801653
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — merestinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NSCLC (Met Exon 14 Mutation) (Experimental): Merestinib at the recommended phase II dose of 120 mg by mouth daily.
  Interventions: Drug: Merestinib
- Solid Tumor (NTRK1,2,3 Rearrangement) (Experimental): Merestinib at the recommended phase II dose of 120 mg by mouth daily.
  Interventions: Drug: Merestinib

INTERVENTIONS:
Drug: Merestinib — Merestinib is a potent and selective type II MET/RON kinase inhibitor with the ability to achieve inhibition of MET activity both in vitro and in vivo.
  Other Names: LY2801653

SUMMARY:
This research study is examining merestinib (a targeted therapy) as a possible treatment for non-small cell lung cancer (NSCLC) that was found to have a specific change in the MET gene (a MET exon 14 mutation); or as a treatment for solid tumors that have an alteration in the NTRK gene (an NTRK1, 2, or 3 rearrangement).

DETAILED DESCRIPTION:
This is an open-label, phase II study of merestinib in patients with advanced NSCLC with a MET exon 14 mutation or patients with advanced cancer harboring an NTRK1, 2, or 3 rearrangement. Twenty patients with a MET mutation will be evaluated in a single-arm design. A small separate cohort of 5 NTRK patients will be evaluated for exploratory purposes.

Merestinib (LY2801653) is a small molecule that has been shown in vitro to be a reversible type II ATP-competitive inhibitor of MET. Pre-clinical testing also has shown merestinib to inhibit several other receptor tyrosine oncokinases including MST1R, FLT3, AXL, MERTK, TEK, ROS1, NTRK1/2/3, and DDR1/2 and the serine/threonine kinases MKNK1/2.

ELIGIBILITY:
Inclusion Criteria:

* Baseline evaluations are to be conducted within 14 days prior to start of protocol therapy, with the exception of the informed consent and baseline tumor imaging which may be obtained up to 28 days prior to the start of protocol therapy.
* For enrollment into the MET cohort: Participants must have a histologically or cytologically confirmed advanced NSCLC and must have received at least one prior line of therapy in the metastatic setting.
* For enrollment into the NTRK cohort: Participants must have a histologically or cytologically confirmed advanced solid tumor and must have received at least one prior line of therapy in the metastatic setting.
* Participants enrolling into the MET cohort must have a MET exon 14 mutation as confirmed by targeted NextGen Sequencing using the DFCI/BWH OncoPanel or another CLIA-certified method. Participants whose NSCLC specimens contain actionable genetic mutations/alterations (e.g. ALK/EGFR) should receive appropriate targeted therapies prior to enrollment in the trial.
* Participants enrolling into the NTRK cohort must have an NTRK1, 2, or 3 rearrangement as confirmed by targeted NextGen Sequencing using the DFCI/BWH OncoPanel or another CLIA-certified method.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Participants enrolling to the MET cohort who have received treatment with a prior MET inhibitor must be able and willing to undergo a baseline tumor biopsy.
* Participants enrolling to the NTRK cohort who have received treatment with a prior NTRK inhibitor must be able and willing to undergo a baseline tumor biopsy.
* Age ≥ 18 years. As no dosing or adverse event data are currently available in participants < 18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* ECOG performance status ≤ 1 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/uL
  * Platelets ≥ 100 K/uL
  * Hemoglobin ≥ 9 g/dL (with or without transfusion support)
  * Total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT)≤ 2.5 × institutional ULN, unless liver metastases are present and then ≤ 5 × institutional ULN is acceptable
  * Serum creatinine ≤ 1.5 × institutional ULN
* The effects of merestinib on the developing human fetus are unknown. For this reason and because MET inhibitor agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of merestinib administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must be able to swallow and retain oral medication or have an enteral feeding tube in place for study drug administration.
* Participants who have received prior oral tyrosine kinase inhibitors (TKIs) will be allowed on study if at least 5 half-lives have elapsed since the date of their last dose of TKI.

Exclusion Criteria:

* Participants who have had chemotherapy, immune therapy, other investigational therapy, major surgery, or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Participants who have not recovered to eligibility levels from adverse events due to agents administered more than 3 weeks earlier.
* Participants who are receiving any other investigational agents.
* Participants with untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Participants with a history of brain metastases that have been treated, are no longer taking corticosteroids, and have been stable on imaging for ≥ 4 weeks following the last date of treatment are permitted. Note: a brain MRI is required during the screening period.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to merestinib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because merestinib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with merestinib, breastfeeding should be discontinued if the mother is treated with merestinib.
* Known HIV-positive participants are ineligible because these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Participants enrolling to the MET cohort who have received a prior MET inhibitor may not be on anticoagulant therapy unless the investigator has deemed it safe to temporarily hold to facilitate the baseline tumor biopsy.
* Participants enrolling to the NTRK cohort who have received a prior NTRK inhibitor may not be on anticoagulant therapy unless the investigator has deemed it safe to temporarily hold to facilitate the baseline tumor biopsy.
* Participants with uncontrolled high blood pressure, defined as a blood pressure during screening of ≥ 160/100 despite medical management.
* Participants must not have any clinically significant gastrointestinal abnormalities that in the opinion of the treating investigator may alter absorption of oral medications, such as malabsorption syndrome or major resection of the stomach or bowels.
* Participants with a history of a second primary malignancy. Exceptions include: patients with a history of malignancies that were treated curatively and have not recurred within 3 years prior to study entry; resected basal and squamous cell carcinomas of the skin, and completely resected carcinoma in situ of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Awad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan SB, Um SL, Peek VL, Stephens JR, Zeng W, Konicek BW, Liu L, Manro JR, Wacheck V, Walgren RA. MET-targeting antibody (emibetuzumab) and kinase inhibitor (merestinib) as single agent or in combination in a cancer model bearing MET exon 14 skipping. Invest New Drugs. 2018 Aug;36(4):536-544. doi: 10.1007/s10637-017-0545-x. Epub 2017 Nov 29. PMID 29188469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between December 2016 to November 2019.
Groups:
- NSCLC (Met Exon 14 Mutation): Merestinib: Oral, predetermined dosage of 120mg per protocol, once daily per 28 day treatment cycle
- Solid Tumor (NTRK1,2,3 Rearrangement): Merestinib: Oral, predetermined dosage of 120 mg per protocol, once daily per 28 day treatment cycle
Period: Overall Study
Arm/Group | NSCLC (Met Exon 14 Mutation) | Solid Tumor (NTRK1,2,3 Rearrangement)
Started | 12 | 0
Completed | 0 | 0
Not Completed | 12 | 0
Not completed — Adverse Event | 8 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Not completed — Missing | 1 | 0
Not completed — Subject Non-Compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patient was accrued in the solid tumor arm.
Groups:
- Solid Tumor (NTRK1,2,3 Rearrangement): Merestinib: Oral, predetermined dosage of 120mg per protocol, once daily per 28 day treatment cycle
- Total: Total of all reporting groups
Arm/Group | NSCLC (Met Exon 14 Mutation) | Solid Tumor (NTRK1,2,3 Rearrangement) | Total
Number analyzed (Participants) | 12 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.13 (5.75) |  | 69.13 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 |  | 9
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  | 1
  Not Hispanic or Latino | 10 |  | 10
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 9 |  | 9
  More than one race | 0 |  | 0
  Unknown or Not Reported | 2 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) - MET Exon 14 Cohort
Description: ORR was defined as the proportion of participants achieving complete response (CR) or partial response (PR) as best response on treatment in MET Exon 14 Cohort based on RECISTv1.1 criteria.
Time Frame: ORR evaluation starting at cycle 2 day 28 and at the end of every 2 cycles of treatment thereafter. The median treatment duration is 1.20 months with range (0.26 months - 28.81 months).
Population: The analysis population is comprised of eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of paticipants
Arm/Group | NSCLC (Met Exon 14 Mutation)
Number analyzed (Participants) | 12
proportion of paticipants | 0.083 [0.002 to 0.4643]

2. Secondary Outcome: Median Overall Survival (OS) - MET Exon 14 Cohort
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Survival data collection in long-term follow-up every 3 months. Median follow-up for survival is of 24.28 months with range (0.46 months - 32.13 months).
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NSCLC (Met Exon 14 Mutation)
Number analyzed (Participants) | 12
months | 24.28 [9.20 to NA] — The upper limit of the 90% CI is not statistically reachable.

3. Secondary Outcome: Median Progression-free Survival (PFS) - MET Exon 14 Cohort
Description: PFS based on the Kaplan-Meier method is defined as the duration between randomization and documented disease progression (PD) defined per RECIST 1.1 criteria. or death, or is censored at time of last disease assessment.
Time Frame: Disease was evaluated at cycle 2 day 28 and at the end of every 2 cycles thereafter and in long-term survival followed-up every 3 months. Median follow-up for survival is of 24.28 months with range (0.46 months - 32.13 months).
Population: The analysis population is comprised of all eligible and treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NSCLC (Met Exon 14 Mutation)
Number analyzed (Participants) | 12
months | 3.68 [1.38 to NA] — There were only 10 events, therefore the upper limit of the 90% CI is not finite.

4. Secondary Outcome: Median Duration of Response (DOR) - MET Exon 14 Cohort
Description: DOR, estimated using the Kaplan Meier method, is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) per RECISTv1.1, until the first date that recurrent or progressive disease is objectively documented. Patients without PD are censored at the date of last disease assessment.
Time Frame: Radiologic evaluation starting at cycle 2 day 28 and at the end of every 2 cycles of treatment thereafter. The median of treatment duration is 1.20 months with range (0.26 months - 28.81 months).
Population: This analysis dataset is comprised of all patients who had a CR or PR on treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | NSCLC (Met Exon 14 Mutation)
Number analyzed (Participants) | 1
months | NA [NA to NA] — Only one patient had a CR/PR on treatment. This study lacks meaningful results and privacy, so the results are unreported.

5. Secondary Outcome: Grade 4-5 Treatment-related Toxicity Rate
Description: All grade 4-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 that are not resolved in accordance with treatment guidelines were counted. Rate is the proportion of treated participants experiencing at least one of these adverse events as defined during the time of observation.
Time Frame: AE evaluated on treatment on day 1 and 15 on cycle 1, and day 1 on each cycle thereafter. The median of treatment duration is 1.20 months with range (0.26 months - 28.81 months).
Population: This analysis dataset is comprised of all eligible and treated patients.
Measure: Number (95% Confidence Interval); unit: proportion of paticipants
Arm/Group | NSCLC (Met Exon 14 Mutation)
Number analyzed (Participants) | 12
proportion of paticipants | 0.083 [0.002 to 0.46]

ADVERSE EVENTS:
Time Frame: AE evaluated on treatment on day 1 and 15 on cycle 1, and day 1 on each cycle thereafter. The median of observation time for AE is 1.20 months with range (0.26 months - 28.81 months). The median of the observation period for all-cause mortality is 24.28 months with range (0.46 months - 32.13 months).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | NSCLC (Met Exon 14 Mutation) | Solid Tumor (NTRK1,2,3 Rearrangement)
All-Cause Mortality (participants affected / at risk) | 7/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/12 | 0/0
Other Adverse Events (participants affected / at risk) | 12/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC (Met Exon 14 Mutation) (N=12) | Solid Tumor (NTRK1,2,3 Rearrangement) (N=0)
Edema limbs (General disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
CPK increased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NSCLC (Met Exon 14 Mutation) (N=12) | Solid Tumor (NTRK1,2,3 Rearrangement) (N=0)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Edema limbs (General disorders) | 5 | 0
Fatigue (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pain (General disorders) | 3 | 0
Alanine aminotransferase increased (Investigations) | 5 | 0
Alkaline phosphatase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 2 | 0
CPK increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 0
Investigations - Other, specify (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT02920996/Prot_SAP_000.pdf